CLINICAL TRIAL: NCT02483988
Title: The SUN Clinical Trial (Safety Utilizing NUsurface Meniscus Implant). A Multi-center, Single-arm, Prospective, Open-label, Non-randomized, Observational Clinical Study
Brief Title: The SUN Clinical Trial (Safety Utilizing NUsurface Meniscus Implant)
Acronym: SUN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Active Implants (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00571
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Post-Meniscectomy Pain Syndrome; Osteoarthritis, Knee
Keywords: NUsurface; Meniscus; prosthesis; KOOS
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- NUsurface Meniscus Implant (Experimental): All eligible patients will receive the NUsurface® Meniscus Implant.
  Interventions: Device: NUsurface® Meniscus Implant

INTERVENTIONS:
Device: NUsurface® Meniscus Implant — The NUsurface® Meniscus Implant is a Polycarbonate-Urethane (PCU)-based device reinforced with high tensile Ultra High Molecular Weight Polyethylene (UHMWPE) fibers. The product is available in different sizes, left and right, and with trials so as to allow the surgeon several size options for implantation. The NUsurface® Meniscus Implant, is designed to be conceptually analogous to the natural meniscus whose structural characteristics include a highly orientated collagen fiber network that supports the large hoop stresses to produce better distribution of contact pressures within the knee joint. Restoring the distribution of joint loads post-meniscectomy is thought to reducing joint overload and to reducing pain.

SUMMARY:
The NUsurface® Meniscus Implant SUN Clinical Trial is a multi-center, single-arm, prospective, open label, non-randomized, observational clinical trial to gather safety and probable clinical benefit data on the NUsurface® Meniscus Implant in treated the target population.

ELIGIBILITY:
Inclusion Criteria:

1. Had > 6 months ago a medial partial meniscectomy as confirmed by patient history and MRI
2. Has a KOOS Pain of ≤ 75 (100 being the highest attainable and no pain)
3. Is between age 30 and 75 years (inclusive) at the time of study treatment
4. Has neutral alignment ±5º of the mechanical axis, as measured from the angle formed by a line drawn from the center of the femoral head to the medial tibial spine and a line drawn from the medial tibial spine and the center of the ankle joint
5. Has ≥ 2 mm intact medial meniscal rim capable of being fitted with a NUsurface® device
6. Is able to do the study required follow-up visits, questionnaires, X-rays and MRI's
7. Is able to read and understand the English language if treated at a U.S. site or read and understand one of the official country languages if treated at a site Outside the U.S.
8. Is able and willing to understand and sign the Informed Consent Form

Exclusion Criteria:

1. Has a symptomatic knee because of a tear that could be addressed by a repeat partial meniscectomy leaving > 4 mm of medial meniscus rim
2. Has evidence of a Outerbridge Grade IV cartilage loss on the medial tibial plateau or femoral condyle that potentially could contact a NUsurface implant (e.g., a focal lesion > 0.5 cm2 correlating to a circular defect of > 8 mm in diameter)
3. Has complete disruption of the posterior root attachment of the meniscus
4. Has lateral compartment pain and Grade III or Grade IV Outerbridge cartilage score in the lateral compartment
5. Has a varus or valgus knee deformity > 5º requiring a tibial or femoral osteotomy
6. Has a laxity level of more than Grade II (IKDC), primary or secondary to an injury of the anterior cruciate ligament (ACL) and/or posterior cruciate ligament (PCL) and/or lateral collateral ligament (LCL) and/or medial collateral ligament (MCL)
7. Has significant trochlear dysplasia, patellar instability or symptomatic patellar misalignment
8. Has patellar compartment pain and Grade III or Grade IV Outerbridge cartilage score in the patellar compartment.
9. Compared to a normal knee, has obvious radiological evidence of medial femoral squaring, anatomical variance in the medial tibial plateau, or irregularly shaped cartilage surface
10. Had an ACL reconstruction performed < 9 months prior to study treatment
11. Has a BMI > 32.5 at the start of study treatment
12. Decides to receive (if eligible and an option) allograft medial meniscus transplantation
13. Received any type of prosthetic knee implant made of artificial non-resorbable plastic, metal or ceramic, not including the NUsurface® Meniscus Implant
14. Has a knee flexion contracture > 10º
15. Has flexion < 90º
16. Had a previous medial femoral condyle surgery (not including microfracture) or High Tibial Osteotomy (HTO)
17. Has insufficiency fractures or avascular necrosis of the medial compartment
18. Has an active infection or tumor (local or systemic)
19. Has any type of knee joint inflammatory disease including Sjogren's syndrome
20. Has neuropathic knee osteoarthropathy, also known as Charcot joint
21. Has any medical condition that does not allow possible arthroscopy of the knee
22. Has neurological deficit (sensory, motor, or reflex)
23. Is currently involved in another investigation of the lower extremity
24. Anticipates having another lower extremity surgery during the study period
25. Is contraindicated for hyaluronic acid injections (i.e., patients with known hypersensitivity [allergy] to hyaluronan [sodium hyaluoronate] preparations); patients having knee joint infections or skin diseases or infections in the site of possible injections
26. Is contraindicated for corticosteroid injections (i.e., patients with allergy to any of the components or with idiopathic thrombocytopenic purpura)
27. Has received any corticosteroid knee injections ≤ 3 months prior to study treatment
28. Has chondrocalcinosis
29. Is on immunostimulating or immunosuppressing agents
30. Has ipsilateral or contralateral lower limb joint conditions that may affect ambulation or KOOS (e.g. have a leg length discrepancy > 2.5 cm [1 inch], causing a noticeable limp)
31. Is a female who is lactating, expecting, or is intending to become pregnant during the study period
32. Is an active smoker
33. Is mentally incapacitated (incapable of appraising or controlling conduct) or have mental disability (e.g., dementia or Alzheimer's)
34. Is a prisoner
35. Is a patient who has economic incentive not to improve
36. Certain patient populations that are at high risk for poor healing or outcomes such as patients who have a co-morbidity that reduces life expectancy to less than 36 months
37. Patients who are contraindicated for MRI (i.e., pacemaker, defibrillator, cochlear implants, etc.)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety assessed by Serious and non-serious, device-related and non-device related adverse events | 2 years
  Safety assessed by Serious and non-serious, device-related and non-device related adverse events recorded during the implantation, up to 24 months following implantation
Clinical Performance | 2 years
  Evaluation of performance defined as NUsurface® Meniscus Implant providing knee pain reduction and improvement in functionality and quality of life up to 24 months post-implantation, as measured by KOOS Pain and KOOS 5

SECONDARY OUTCOMES:
Safety assessed by Serious and non-serious, device-related and non-device related adverse events | 5 years
  Safety assessed by Serious and non-serious, device-related and non-device related adverse events occurring between 24 and 60 months following implantation
Clinical Performance | 5 years
  Evaluation of performance defined as NUsurface® Meniscus Implant providing knee pain reduction and improvement in functionality and quality of life up to 60 months post-implantation, as measured by KOOS Pain and KOOS 5

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Treharne, PhD, Study Director — Active Implants LLC
Locations (13):
- United States (13):
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Horizon Clinical Research, La Mesa, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - St Mary's Medical Center, San Francisco, California
  - CU Sports Medicine, Boulder, Colorado
  - Advanced Orthopaedics & Sports Medicine Specialists, Denver, Colorado
  - OrthoIndy, Greenwood, Indiana
  - Baton Rouge Orthopaedic Clinic, Baton Rouge, Louisiana
  - Ochsner Sports Medicine Institute, New Orleans, Louisiana
  - Sports Medicine Oregon, Portland, Oregon
  - Arlington Orthopedic Associates, PA, Arlington, Texas
  - Comprehensive Orthopaedics & Sports Medicine, Salt Lake City, Utah
  - OrthoVirginia, Richmond, Virginia

REFERENCES:
- [Background] De Coninck T, Elsner JJ, Linder-Ganz E, Cromheecke M, Shemesh M, Huysse W, Verdonk R, Verstraete K, Verdonk P. In-vivo evaluation of the kinematic behavior of an artificial medial meniscus implant: A pilot study using open-MRI. Clin Biomech (Bristol). 2014 Sep;29(8):898-905. doi: 10.1016/j.clinbiomech.2014.07.001. Epub 2014 Jul 17. PMID 25238685
- [Background] Shemesh M, Asher R, Zylberberg E, Guilak F, Linder-Ganz E, Elsner JJ. Viscoelastic properties of a synthetic meniscus implant. J Mech Behav Biomed Mater. 2014 Jan;29:42-55. doi: 10.1016/j.jmbbm.2013.08.021. Epub 2013 Sep 3. PMID 24055793
- [Background] Zur G, Linder-Ganz E, Elsner JJ, Shani J, Brenner O, Agar G, Hershman EB, Arnoczky SP, Guilak F, Shterling A. Chondroprotective effects of a polycarbonate-urethane meniscal implant: histopathological results in a sheep model. Knee Surg Sports Traumatol Arthrosc. 2011 Feb;19(2):255-63. doi: 10.1007/s00167-010-1210-5. Epub 2010 Jul 16. PMID 20635076
- [Background] Elsner JJ, Portnoy S, Guilak F, Shterling A, Linder-Ganz E. MRI-based characterization of bone anatomy in the human knee for size matching of a medial meniscal implant. J Biomech Eng. 2010 Oct;132(10):101008. doi: 10.1115/1.4002490. PMID 20887018
- [Background] Elsner JJ, Portnoy S, Zur G, Guilak F, Shterling A, Linder-Ganz E. Design of a free-floating polycarbonate-urethane meniscal implant using finite element modeling and experimental validation. J Biomech Eng. 2010 Sep;132(9):095001. doi: 10.1115/1.4001892. PMID 20815651
- [Background] Linder-Ganz E, Elsner JJ, Danino A, Guilak F, Shterling A. A novel quantitative approach for evaluating contact mechanics of meniscal replacements. J Biomech Eng. 2010 Feb;132(2):024501. doi: 10.1115/1.4000407. PMID 20370247
- [Background] Elsner JJ, Shemesh M, Shefy-Peleg A, Gabet Y, Zylberberg E, Linder-Ganz E. Quantification of in vitro wear of a synthetic meniscus implant using gravimetric and micro-CT measurements. J Mech Behav Biomed Mater. 2015 Sep;49:310-20. doi: 10.1016/j.jmbbm.2015.05.017. Epub 2015 May 28. PMID 26057364